CLINICAL TRIAL: NCT02575352
Title: Observational Prospective Multi-center International Study on the Use of Injectable Calcium Phosphate Cements for the Treatment of Bone Defects in Adults.
Brief Title: Calcium Phosphate Cement Registry (CPC Registry)
Acronym: CPC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Graftys SA (Industry)
Collaborators: Clinfile (Industry)
Responsible Party: Sponsor
Other Study IDs: GR-NI-INJ
Record Dates: First submitted 2015-10-12; First posted 2015-10-14 (Estimated); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Bone Disease; Fracture Bone; Bone Cyst
Keywords: Bone Substitute; Calcium Phosphate Cement; GRAFTYS; GRAFTYS®HBS; GRAFTYS®QUICKSET; Bone void filler; Bone growth; Registry; Bone defect; Revision arthroplasty; Arthrodesis
MeSH Terms: conditions — Bone Diseases; Fractures, Bone; Bone Cysts; Ankylosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
CPC REGISTRY is a multi-center, international, prospective, open-label, observational study on the use of injectable calcium phosphate cements for the treatment of bone defects in adults. All patients will be treated with any of the two injectable calcium phosphate bone substitutes (GRAFTYS®HBS/GRAFTYS®Quickset or their private labels) according to standard clinical practice and according to the information provided by GRAFTYS manufacturer in respective device Instructions For Use (IFU).

DETAILED DESCRIPTION:
The objective of this observational prospective study is to collect safety and performance data relating to the use of injectable Calcium Phosphate Cements "GRAFTYS®HBS/GRAFTYS®Quickset (or their private labels)" in routine clinical practice from various international hospitals. Therefore this observational study will allow to support data about risk management (established at the end of the product development); and to enhance the current clinical evaluation of products with new clinical data (for longer follow-up). The collected data of this observational study will be "non-identifying data". The patient must have signed a Written Consent Form (for data collection) prior to any data being entered into the electronic Case Report Form.

Patients will be followed as per local standard medical practices of the center for two years. Five follow-up visits/phone calls will be collected (at 3 months (+/-14 days), 6 months (+/- 14 days), 9 months (+/-21 days), 12 months (+/- 30 days) and 24 months (+/-60 days)). Each visit/phone call includes the collection of Adverse Events, the measurement of health status (quality of life and functional scores) and the X-ray scoring (if X-ray imaging is available). No additional exams (other than the routine clinical practice) are requested. The surgeons have to follow their usual practices (e.g. X-Rays have to be performed only if they are scheduled in the routine clinical practice).

All Adverse Events will be collected and monitored at each follow-up visit or follow-up phone call. All Serious Adverse Events must be described via a Serious Adverse Event form in e-CRF and all Adverse Device Effects must be described via a "Product Complaint Form" in e-CRF.

Descriptive analyses will be performed in order to describe: nature of adverse events, their distribution and frequency. Moreover, all factors which may appear predictive for the rate of adverse events will be analyzed (age, sex, amount of CPC injected, delivery system used, diabetes history, smoking habits, alcohol consumption, concomitant treatments/diseases…). For all time-dependent events, life-tables will be able to calculate using the Kaplan Meier estimate method, for a period starting on the date of the procedure up to and including the 24-months follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Bone skeletal defects that are not intrinsic to the stability of bone structure OR site which can be stabilized
2. Bone defects from surgery, trauma, tumor or cyst
3. Age ≥ 18 years
4. Patient information and signed informed consent form (for data collection)
5. Affiliation to a Social Security System schema (or similar system)

Exclusion Criteria:

1. Patients undergoing radiotherapy or chemotherapy
2. Patients with inflammatory bone disease
3. Patients with a calcium metabolism anomaly, severe metabolic disease, vascular or neurological diseases, or immunological deficiencies
4. Bone site which can lead to the product passing into the joint cavities without appropriate controls (visual, arthroscopic, lavage…).
5. Bone site which can lead to the product passing into the meningeal spaces
6. Vertebroplasty and kyphoplasty
7. Site infected or one suspected of being so
8. A cranio-maxillofacial defect with a surface area larger than 25 cm2
9. A site exposed to the sinus (lumen) or nasal mucosa
10. Pregnant women (or likely to be) or breast-feeding women
11. Inability to understand the consent and objectives of the study
12. Unable to undergo medical monitoring for geographical, social or psychological reasons
13. Persons who are deprived of liberty or under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients eligible and planned for bone defect treatment who meet predefined criteria in Instructions For Use (IFU) of GRAFTYS®HBS/ GRAFTYS®Quickset.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-05 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Adverse Device Effect rate | For 24 months
  Rate of Adverse Events related to bone substitutes (registry devices) for the follow-up period of patients.

SECONDARY OUTCOMES:
Technical Success rate | At surgical procedure
  Technical Success rate defined as successful delivery of the bone substitute in the target defect bone without evidence of delivery device or bone substitute malfunction. (NOTE: Malfunction is definied as a failure of the medical device to perform in accordance with its intended purpose when used in accordance with the Instructions For Uses (IFU)).
Device Deficiencies rate | At surgical procedure
  Device deficiency is defined as an inadequacy of a medical device with respect to its identity, quality, durability, reliability, safety or performance.
  NOTE: Device deficiencies include malfunctions, use errors, and inadequate labelling.
Serious Adverse Events rate in the peroperative period | At surgical procedure
  Serious Adverse Event is defined as any adverse event that:
  1. Led to a death,
  2. Led to serious deterioration in health of the subject that either resulted in:
     1. a life-threatening illness or injury, or
     2. a permanent impairment of a body structure or a body function, or
     3. in-patient or prolonged hospitalization, or
     4. medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function.
  3. Led to fetal distress, fetal death or a congenital abnormality or birth defect.
Serious Adverse Events rate during the follow-up period | 3 months post index procedure
  Serious Adverse Event is defined as any adverse event that:
  1. Led to a death,
  2. Led to serious deterioration in health of the subject that either resulted in:
     1. a life-threatening illness or injury, or
     2. a permanent impairment of a body structure or a body function, or
     3. in-patient or prolonged hospitalization, or
     4. medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function.
  3. Led to fetal distress, fetal death or a congenital abnormality or birth defect.
Serious Adverse Events rate during the follow-up period | 6 months post index procedure
  Serious Adverse Event is defined as any adverse event that:
  1. Led to a death,
  2. Led to serious deterioration in health of the subject that either resulted in:
     1. a life-threatening illness or injury, or
     2. a permanent impairment of a body structure or a body function, or
     3. in-patient or prolonged hospitalization, or
     4. medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function.
  3. Led to fetal distress, fetal death or a congenital abnormality or birth defect.
Serious Adverse Events rate during the follow-up period | 9 months post index procedure
  Serious Adverse Event is defined as any adverse event that:
  1. Led to a death,
  2. Led to serious deterioration in health of the subject that either resulted in:
     1. a life-threatening illness or injury, or
     2. a permanent impairment of a body structure or a body function, or
     3. in-patient or prolonged hospitalization, or
     4. medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function.
  3. Led to fetal distress, fetal death or a congenital abnormality or birth defect.
Serious Adverse Events rate during the follow-up period | 12 months post index procedure
  Serious Adverse Event is defined as any adverse event that:
  1. Led to a death,
  2. Led to serious deterioration in health of the subject that either resulted in:
     1. a life-threatening illness or injury, or
     2. a permanent impairment of a body structure or a body function, or
     3. in-patient or prolonged hospitalization, or
     4. medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function.
  3. Led to fetal distress, fetal death or a congenital abnormality or birth defect.
Serious Adverse Events rate during the follow-up period | 24 months post index procedure
  Serious Adverse Event is defined as any adverse event that:
  1. Led to a death,
  2. Led to serious deterioration in health of the subject that either resulted in:
     1. a life-threatening illness or injury, or
     2. a permanent impairment of a body structure or a body function, or
     3. in-patient or prolonged hospitalization, or
     4. medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function.
  3. Led to fetal distress, fetal death or a congenital abnormality or birth defect.
Bone reconstruction evolution after surgery (if X-rays are available) | 3 months post index procedure
  X-ray scoring systems have been implemented according to the medical literature criteria. For trauma defects/arthrodesis, the results are scored using the criteria proposed by Lane and Sandhu (bone formation, union and remodeling) and also including a bone substitute resorption (radiolucency) criteria. As for prosthesis revision/cavity defects, the scoring system includes bone substitute resorption, bone formation, remodeling and presence or absence of a radiolucent line between the bone and the cement/implant. The maximum score for both groups (trauma/arthrodesis & cavity filling/arthroplasty) is 10/10 (excellent consolidation/excellent secondary stabilization) and the minimum score is 0/10 (no consolidation/no secondary stabilization).
Bone reconstruction evolution after surgery (if X-rays are available) | 6 months post index procedure
  X-ray scoring systems have been implemented according to the medical literature criteria. For trauma defects/arthrodesis, the results are scored using the criteria proposed by Lane and Sandhu (bone formation, union and remodeling) and also including a bone substitute resorption (radiolucency) criteria. As for prosthesis revision/cavity defects, the scoring system includes bone substitute resorption, bone formation, remodeling and presence or absence of a radiolucent line between the bone and the cement/implant. The maximum score for both groups (trauma/arthrodesis & cavity filling/arthroplasty) is 10/10 (excellent consolidation/excellent secondary stabilization) and the minimum score is 0/10 (no consolidation/no secondary stabilization).
Bone reconstruction evolution after surgery (if X-rays are available) | 9 months post index procedure
  X-ray scoring systems have been implemented according to the medical literature criteria. For trauma defects/arthrodesis, the results are scored using the criteria proposed by Lane and Sandhu (bone formation, union and remodeling) and also including a bone substitute resorption (radiolucency) criteria. As for prosthesis revision/cavity defects, the scoring system includes bone substitute resorption, bone formation, remodeling and presence or absence of a radiolucent line between the bone and the cement/implant. The maximum score for both groups (trauma/arthrodesis & cavity filling/arthroplasty) is 10/10 (excellent consolidation/excellent secondary stabilization) and the minimum score is 0/10 (no consolidation/no secondary stabilization).
Bone reconstruction evolution after surgery (if X-rays are available) | 12 months post index procedure
  X-ray scoring systems have been implemented according to the medical literature criteria. For trauma defects/arthrodesis, the results are scored using the criteria proposed by Lane and Sandhu (bone formation, union and remodeling) and also including a bone substitute resorption (radiolucency) criteria. As for prosthesis revision/cavity defects, the scoring system includes bone substitute resorption, bone formation, remodeling and presence or absence of a radiolucent line between the bone and the cement/implant. The maximum score for both groups (trauma/arthrodesis & cavity filling/arthroplasty) is 10/10 (excellent consolidation/excellent secondary stabilization) and the minimum score is 0/10 (no consolidation/no secondary stabilization).
Bone reconstruction evolution after surgery (if X-rays are available) | 24 months post index procedure
  X-ray scoring systems have been implemented according to the medical literature criteria. For trauma defects/arthrodesis, the results are scored using the criteria proposed by Lane and Sandhu (bone formation, union and remodeling) and also including a bone substitute resorption (radiolucency) criteria. As for prosthesis revision/cavity defects, the scoring system includes bone substitute resorption, bone formation, remodeling and presence or absence of a radiolucent line between the bone and the cement/implant. The maximum score for both groups (trauma/arthrodesis & cavity filling/arthroplasty) is 10/10 (excellent consolidation/excellent secondary stabilization) and the minimum score is 0/10 (no consolidation/no secondary stabilization).
Quality of life score at baseline (EQ-5D-3L) | At baseline (pre-operative)
  This health status information is collected before and after a procedure and provides an indication of the clinical outcomes or quality of care delivered to patients. EQ-5D-3L paper questionnaire will be self-administered or it will be administered to patient via a telephone interview. The EQ-5D-5L still consists of 2 parts - the EQ-5D-5L descriptive system and the EQ VAS. The descriptive system comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression). Each dimension has 3 levels: no problems, some problems, extreme problems. EQ VAS is a scale on which the "best imaginable health state" is marked 100 and the "worst imaginable state" is marked 0.
Quality of life score evolution after surgery (EQ-5D-3L) | 3 months post index procedure
  This health status information is collected before and after a procedure and provides an indication of the clinical outcomes or quality of care delivered to patients. EQ-5D-3L paper questionnaire will be self-administered or it will be administered to patient via a telephone interview. The EQ-5D-5L still consists of 2 parts - the EQ-5D-5L descriptive system and the EQ VAS. The descriptive system comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression). Each dimension has 3 levels: no problems, some problems, extreme problems. EQ VAS is a scale on which the "best imaginable health state" is marked 100 and the "worst imaginable state" is marked 0.
Quality of life score evolution after surgery (EQ-5D-3L) | 6 months post index procedure
  This health status information is collected before and after a procedure and provides an indication of the clinical outcomes or quality of care delivered to patients. EQ-5D-3L paper questionnaire will be self-administered or it will be administered to patient via a telephone interview. The EQ-5D-5L still consists of 2 parts - the EQ-5D-5L descriptive system and the EQ VAS. The descriptive system comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression). Each dimension has 3 levels: no problems, some problems, extreme problems. EQ VAS is a scale on which the "best imaginable health state" is marked 100 and the "worst imaginable state" is marked 0.
Quality of life score evolution after surgery (EQ-5D-3L) | 9 months post index procedure
  This health status information is collected before and after a procedure and provides an indication of the clinical outcomes or quality of care delivered to patients. EQ-5D-3L paper questionnaire will be self-administered or it will be administered to patient via a telephone interview. The EQ-5D-5L still consists of 2 parts - the EQ-5D-5L descriptive system and the EQ VAS. The descriptive system comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression). Each dimension has 3 levels: no problems, some problems, extreme problems. EQ VAS is a scale on which the "best imaginable health state" is marked 100 and the "worst imaginable state" is marked 0.
Quality of life score evolution after surgery (EQ-5D-3L) | 12 months post index procedure
  This health status information is collected before and after a procedure and provides an indication of the clinical outcomes or quality of care delivered to patients. EQ-5D-3L paper questionnaire will be self-administered or it will be administered to patient via a telephone interview. The EQ-5D-5L still consists of 2 parts - the EQ-5D-5L descriptive system and the EQ VAS. The descriptive system comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression). Each dimension has 3 levels: no problems, some problems, extreme problems. EQ VAS is a scale on which the "best imaginable health state" is marked 100 and the "worst imaginable state" is marked 0.
Quality of life score evolution after surgery (EQ-5D-3L) | 24 months post index procedure
  This health status information is collected before and after a procedure and provides an indication of the clinical outcomes or quality of care delivered to patients. EQ-5D-3L paper questionnaire will be self-administered or it will be administered to patient via a telephone interview. The EQ-5D-5L still consists of 2 parts - the EQ-5D-5L descriptive system and the EQ VAS. The descriptive system comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression). Each dimension has 3 levels: no problems, some problems, extreme problems. EQ VAS is a scale on which the "best imaginable health state" is marked 100 and the "worst imaginable state" is marked 0.
Functional score at baseline (if applicable according to the type of bone defect/medical indication). | At baseline (pre-operative)
  Functional scores are used to monitor the patient progress. The questionnaires concern the degree of difficulty (level of function) that the patient experienced in performing usual daily activities and higher level activities due to his bone defect. Therefore, the type of functional score depends on the skeletal region impacted by the bone defect:
  * Hand/wrist/ elbow/shoulder: Quick-DASH score (Disabilities of Arm, Shoulder & Hand).
  * Knee: KOOS-PS (Knee Injury & Osteoarthritis Outcome Score- Physical function Short form)
  * Hip: HOOS-PS (Hip disability and Osteoarthritis Outcome Score- Physical function Short form)
  * Foot/Ankle: Kitaoka & al's criteria, AOFAS Ankle-Hindfoot Scale; Forefoot Scale; Midfoot scale.
Functional score evolution after surgery (if applicable according to the type of bone defect/medical indication). | 3 months post index procedure
  Functional scores are used to monitor the patient progress. The questionnaires concern the degree of difficulty (level of function) that the patient experienced in performing usual daily activities and higher level activities due to his bone defect. Therefore, the type of functional score depends on the skeletal region impacted by the bone defect:
  * Hand/wrist/ elbow/shoulder: Quick-DASH score (Disabilities of Arm, Shoulder & Hand).
  * Knee: KOOS-PS (Knee Injury & Osteoarthritis Outcome Score- Physical function Short form)
  * Hip: HOOS-PS (Hip disability and Osteoarthritis Outcome Score- Physical function Short form)
  * Foot/Ankle: Kitaoka & al's criteria, AOFAS Ankle-Hindfoot Scale; Forefoot Scale; Midfoot scale.
Functional score evolution after surgery (if applicable according to the type of bone defect/medical indication). | 6 months post index procedure
  Functional scores are used to monitor the patient progress. The questionnaires concern the degree of difficulty (level of function) that the patient experienced in performing usual daily activities and higher level activities due to his bone defect. Therefore, the type of functional score depends on the skeletal region impacted by the bone defect:
  * Hand/wrist/ elbow/shoulder: Quick-DASH score (Disabilities of Arm, Shoulder & Hand).
  * Knee: KOOS-PS (Knee Injury & Osteoarthritis Outcome Score- Physical function Short form)
  * Hip: HOOS-PS (Hip disability and Osteoarthritis Outcome Score- Physical function Short form)
  * Foot/Ankle: Kitaoka & al's criteria, AOFAS Ankle-Hindfoot Scale; Forefoot Scale; Midfoot scale.
Functional score evolution after surgery (if applicable according to the type of bone defect/medical indication). | 9 months post index procedure
  Functional scores are used to monitor the patient progress. The questionnaires concern the degree of difficulty (level of function) that the patient experienced in performing usual daily activities and higher level activities due to his bone defect. Therefore, the type of functional score depends on the skeletal region impacted by the bone defect:
  * Hand/wrist/ elbow/shoulder: Quick-DASH score (Disabilities of Arm, Shoulder & Hand).
  * Knee: KOOS-PS (Knee Injury & Osteoarthritis Outcome Score- Physical function Short form)
  * Hip: HOOS-PS (Hip disability and Osteoarthritis Outcome Score- Physical function Short form)
  * Foot/Ankle: Kitaoka & al's criteria, AOFAS Ankle-Hindfoot Scale; Forefoot Scale; Midfoot scale.
Functional score evolution after surgery (if applicable according to the type of bone defect/medical indication). | 12 months post index procedure
  Functional scores are used to monitor the patient progress. The questionnaires concern the degree of difficulty (level of function) that the patient experienced in performing usual daily activities and higher level activities due to his bone defect. Therefore, the type of functional score depends on the skeletal region impacted by the bone defect:
  * Hand/wrist/ elbow/shoulder: Quick-DASH score (Disabilities of Arm, Shoulder & Hand).
  * Knee: KOOS-PS (Knee Injury & Osteoarthritis Outcome Score- Physical function Short form)
  * Hip: HOOS-PS (Hip disability and Osteoarthritis Outcome Score- Physical function Short form)
  * Foot/Ankle: Kitaoka & al's criteria, AOFAS Ankle-Hindfoot Scale; Forefoot Scale; Midfoot scale.
Functional score evolution after surgery (if applicable according to the type of bone defect/medical indication). | 24 months post index procedure
  Functional scores are used to monitor the patient progress. The questionnaires concern the degree of difficulty (level of function) that the patient experienced in performing usual daily activities and higher level activities due to his bone defect. Therefore, the type of functional score depends on the skeletal region impacted by the bone defect:
  * Hand/wrist/ elbow/shoulder: Quick-DASH score (Disabilities of Arm, Shoulder & Hand).
  * Knee: KOOS-PS (Knee Injury & Osteoarthritis Outcome Score- Physical function Short form)
  * Hip: HOOS-PS (Hip disability and Osteoarthritis Outcome Score- Physical function Short form)
  * Foot/Ankle: Kitaoka & al's criteria, AOFAS Ankle-Hindfoot Scale; Forefoot Scale; Midfoot scale.
Surgeon's Satisfaction survey with registry device | At surgical procedure
  Surgeon's Satisfaction survey with registry device (about mixing ability, injecting ability and moldability) thanks to a 100-mm Visual Analog Scale (VAS). A score of zero indicated absolutely inacceptable, while a score of 100 indicated very satisfying.

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien PARRATTE, MD, Prof, Principal Investigator — Hospital of "LA TIMONE"
Locations (11):
- France (4):
  - Hôpital La Timone, Marseille
  - Marseille
  - Paris
  - Saint-Louis
- Germany (3):
  - Kiel
  - Ratzeburg
  - Würzburg
- Italy (2):
  - Palermo
  - Piacenza
- Fort-de-France, Martinique
- Yverdon-les-Bains, Switzerland